CLINICAL TRIAL: NCT05452421
Title: Plasma and Salivary Nitrate/Nitrite Responses and Power Output Compared After Two Beetroot Juice Drinks
Brief Title: Nitrate and Power Output After Two Beetroot Juice Drinks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanyang Technological University (Other)
Responsible Party: Principal Investigator, Stephen Burns, Associate Professor, Nanyang Technological University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: IRB-2022-149
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Blood Plasma Nitrite

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Two drinks similar in colour and texture have been provided by a local manufacturer which are coded. The code is held with a third party not involved in the research. Participants and researchers will be asked to guess which drink has been used at the end of each trial to confirm the effectiveness of the masking procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Isotonic carbohydrate beetroot juice drink
  Interventions: Dietary Supplement: Isotonic carbohydrate beetroot juice drink; Dietary Supplement: Beetroot juice drink
- Group B (Experimental): Beetroot juice drink
  Interventions: Dietary Supplement: Isotonic carbohydrate beetroot juice drink; Dietary Supplement: Beetroot juice drink

INTERVENTIONS:
Dietary Supplement: Isotonic carbohydrate beetroot juice drink — An isotonic carbohydrate beetroot juice drink containing 141 mg nitrate per 100 ml (12.9 mmol). Total of 570 ml serving in two doses of 285 ml over one morning. Contains 6.2 g carbohydrate per 100 ml. Osmolality 304-310 mOsm/kg.
  Other Names: ISO-CB
Dietary Supplement: Beetroot juice drink — A beetroot juice drink containing 141 mg nitrate per 100 ml (12.9 mmol). Total of 570 ml serving in two doses of 285 ml over one morning. Contains 6.1 g carbohydrate per 100 ml. Osmolality 390-410 mOsm/kg.
  Other Names: BR

SUMMARY:
The main aim of this study is to determine and compare the optimal time to achieve peak concentration of blood plasma nitrite after ingestion of beetroot juice (BR) and isotonic beetroot juice (ISO-CB), respectively. Optimal timing of drink consumption in relation to exercise can then be prescribed in relation to nitrite appearance in the blood. A randomised controlled trial with participants completing two conditions: (i) BR and (ii) ISO-CB. On each condition participants will consume During each trial, participants will ingest 2 x 285ml of beverage 3 hours prior to performing two jump tests follow by a Wingate test. Salivary NO content will be measured at the start of the morning, 1 hour, 2 hours, 3 hours after consumption of beverage and at the end of the exercise.

DETAILED DESCRIPTION:
1. The main aim of this study is to determine and compare the optimal time to achieve peak concentration of blood plasma nitrite after ingestion of beetroot juice (BR) and isotonic beetroot juice (ISO-CB), respectively. Optimal timing of drink consumption in relation to exercise can then be prescribed in relation to nitrite appearance in the blood.
2. A secondary aim of this study is to evaluate the association between blood plasma nitrite concentration and saliva nitrite concentration after ingestion of the two drinks to determine whether blood plasma analysis can be fully or partially substituted with a salivary nitrite test.
3. A final aim of this study is to investigate the ergogenic effects of ISO-CB compared with BR during a single 30 second cycling sprint bout (Wingate test) and two jumping tests.

A randomised controlled trial recruiting 24 healthy male and female participants. Each participant will complete two conditions: (i) BR and (ii) ISO-CB. On each condition participants will consume During each trial, participants will ingest 2 x 285ml of beverage 3 hours prior to performing two jump tests follow by a Wingate test. In the next trial, participants will undergo the same procedures, but ingest the beverage that they did not take the previous round. The study will be double-blinded study. Blood samples will be taken before supplementation, 2 hours and 3 hours after consuming the beverage. Salivary NO content will be measured at the start of the morning, 1 hour, 2 hours, 3 hours after consumption of beverage and at the end of the exercise. For each trial, participants will also fill out a sensory evaluation form in relation to the drink consumed. It is hypothesized that blood plasma nitrite and saliva nitrite appearance will be earlier with ISO-CB and that participants will have improved peak and mean power when ISO-CB is consumed compared with BR.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 21-35 years.
2. Healthy and injury-free: defined as no positive (Yes) answers to the Physical Activity Readiness Questionnaire (PAR-Q+) and not reporting any other health issues that may be affected by exercise.
3. Blood pressure: <130/90 mmHg.
4. Physically active: Engaging in a minimum of 150 minutes of moderate-intensity exercise or 75 minutes of vigorous-intensity physical activity each week determined via self-report Global Physical Activity Questionnaire (GPAQ).
5. Body mass index (BMI): 18.5-25.0 kg/m2.
6. Non-smoker.

Exclusion Criteria:

1. Any allergies to beetroot or isotonic drink.
2. Asthma.
3. Any report of personal health issues that may compromise the individual's ability to undertake exercise safely.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Blood plasma nitrite | 3 hours
  Peak concentration of blood plasma nitrite

SECONDARY OUTCOMES:
Salivary nitrite | 3 hours
  Salivary nitrite concentration
Power output | 30 seconds
  Peak and mean power output
Jump height and distance | Two jumps averaged
  Jump height and distance

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Burns, PhD, Principal Investigator — Nanyang Technological University
Locations (1):
- Human Bioenergetics Laboratory, National Institute of Education, Nanyang Technological University, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No